CLINICAL TRIAL: NCT06105775
Title: Inorganic Nitrate Supplementation for Blood Pressure Control in Chronic Hypertensive Pregnancies From the 2nd Trimester (NIT_CH): a Triple-Blind Randomized Placebo-Controlled Trial
Brief Title: Inorganic Nitrate Supplementation in Chronic Hypertensive Pregnancies
Acronym: NIT_CH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Hospital das Clínicas de Ribeirão Preto (Other)
Responsible Party: Principal Investigator, Ricardo de Carvalho Cavalli, Professor Dr, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 21/12010-7-SP2
Record Dates: First submitted 2023-10-23; First posted 2023-10-30 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Hypertension in Pregnancy; Hypertension; Pregnancy
Keywords: Endothelial Dysfunction; Hypertension in Pregnancy; Nitric Oxide; inorganic nitrate
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inorganic Nitrate Capsule (Experimental): Once daily capsule containing sodium nitrate (400 mg of nitrate and 140 mg of sodium), for 154 consecutive days.
  Interventions: Dietary Supplement: Inorganic Nitrate Capsule
- Placebo Capsule. (Placebo Comparator): Once daily capsule containing sodium chloride (140 mg of sodium chloride and 400 mg of flour), for 154 consecutive days.
  Interventions: Dietary Supplement: Placebo Capsule

INTERVENTIONS:
Dietary Supplement: Inorganic Nitrate Capsule — Starting from the 16th week of gestation and continuing for 22 weeks (154 days) or until delivery, whichever comes first, participants will consume a daily capsule containing 400 mg of inorganic nitrate. Participants will maintain standard preeclampsia prophylaxis (acetylsalicylic acid 100mg nightly until 36 weeks of gestation and calcium carbonate 1000mg daily until delivery) and regular antihypertensive treatment.
  Arms: Inorganic Nitrate Capsule
Dietary Supplement: Placebo Capsule — From the 16th week of gestation and lasting 22 weeks (154 days) or until delivery, participants will consume a daily capsule containing sodium chloride with the nitrate replaced by plant-based flour, design to mimic the appearance of the active capsule. Participants will maintain standard preeclampsia prophylaxis (acetylsalicylic acid 100mg nightly until 36 weeks of gestation and calcium carbonate 1000mg daily until delivery) and regular antihypertensive treatment.
  Arms: Placebo Capsule.

SUMMARY:
High blood pressure during pregnancy poses significant risks to both the mother and baby. A combination of factors, including advancing maternal age, rising obesity rates, and metabolic health issues, have amplified the prevalence of this condition. While conventional medicines are available, safety during pregnancy remains a concern. Recent studies suggest that inorganic nitrate might be a safer alternative. The power of nitrate lies in its ability to stimulate the body's production of a compound that aids in dilating and relaxing blood vessels. Preliminary studies conducted on mice and a select group of pregnant women have yielded encouraging results. Early tests indicated that after consuming inorganic nitrate, there was a reduction in blood pressure and an improvement in the health of the mother's uterine artery-a vital vessel responsible for nourishing the fetus. Our study aims to investigate the effects of inorganic nitrate supplementation on pregnant women from the start of their pregnancy and continuing it throughout their term. If our findings are positive, it could revolutionize how we approach blood pressure management during pregnancy, paving the way for healthier futures for both mothers and babies.

DETAILED DESCRIPTION:
Eligible pregnant women with chronic hypertension will be identified and invited to participate through posters displayed in the municipality's health units, as well as by medical professionals within the local health network, based on the inclusion criteria. An appointment will be promptly scheduled to verify eligibility and present the informed consent form, during which all questions and concerns will be addressed.

On the enrollment day, the subsequent visit will be scheduled for the 16th week of their pregnancy, marking the commencement of the study. By then, participants will already have been randomly allocated to respective groups by an external professional who is not directly involved in the study, ensuring blinding. Randomization will occur on a 1:1 ratio, employing blocks of 2-4 pregnant women as determined by specialized software. Regardless of allocation, participants will continue with standard medications for preeclampsia prophylaxis: acetylsalicylic acid, taken at 100 mg nightly up to 36 weeks of gestation, and calcium carbonate, taken at 1000 mg daily until delivery, alongside routine antihypertensive treatment.

From the 16th week of pregnancy onward, participants will receive either a capsule containing 400 mg of inorganic nitrate (540 mg of sodium nitrate, equivalent to 140 mg of sodium chloride and 400 mg of nitrate) or a placebo (140 mg of sodium chloride and 400 mg of flour). Both capsules will be identical in color and appearance. All participants will be instructed to take one capsule each morning, continuing this regimen for 22 weeks (154 days), ending either at the 38th week of pregnancy or at childbirth, whichever occurs first.

Visits will take place at predetermined intervals based on the progression of the pregnancy. Initially set at a frequency of every 4 weeks, but as the end of the pregnancy approaches, the visits will become more frequent. The baseline appointment is set for the 16th week of gestation, with subsequent appointments scheduled for the 20th, 24th, 28th, 32nd, 34th, 36th, 37th, and 38th weeks. It is important to note that scheduled visits may conclude earlier if childbirth occurs sooner, or they might be extended if the pregnancy progresses beyond the anticipated delivery date. During these visits, participants will undergo an obstetric clinical examination, blood pressure measurement, biochemical analysis, and an ultrasound paired with a Doppler study of the uterine arteries.

To ensure consistent and optimal blood pressure levels, the overseeing medical team will closely monitor and adjust participants' antihypertensive medications as necessary. Ensuring adherence to the regimen is paramount; thus, participants will be asked to return any unused capsules during their visits and will then be supplied with their next batch for the ensuing period.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women diagnosed with chronic hypertension (systolic blood pressure above 140 mmHg and/or diastolic blood pressure above 90 mmHg before pregnancy or before 20 weeks of gestation) as defined by the Brazilian Network for Studies on Hypertension in Pregnancy (RBEHG, Brazilian acronym) Protocol and Chronic Hypertension/Preeclampsia by the Brazilian Federation of Gynecology and Obstetrics Associations (FEBRASGO, Brazilian acronym) Protocol.
* Patients on monotherapy with methyldopa as treatment at the time of inclusion.
* Women with less than 16 weeks of gestation confirmed by first-trimester ultrasonography confirming gestational age.

Exclusion Criteria:

* Multiple pregnancies, age below 16 years old, inability to provide informed consent, or history of low adherence to medication therapy.
* Patients with uncontrolled chronic hypertension, with blood pressure values above 160x110mmHg.
* History of food allergies, especially hypersensitivity to beetroot.
* Users of illicit drugs, smokers, or alcohol abusers.
* Diagnosis of coronary artery disease, congestive heart failure (moderate to severe), moderate to severe liver failure, chronic renal insufficiency (with plasma creatinine clearance less than 30 ml/min/1.73 m² of body surface), pre-existing type 1 diabetes, and type 2 diabetes.
* Pregnant women who frequently used non-steroidal anti-inflammatory drugs, nasal decongestants, and anorectics before getting pregnant; users of proton pump inhibitors and H2 receptor antagonists or any other medication that interferes with stomach pH, starting 2 weeks before the beginning and continuing throughout the remainder of the study.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-03-06 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure Control in Chronic Hypertensive Pregnant Women with Inorganic Nitrate Supplementation Compared to Placebo. | From baseline (16th week) up to delivery
  Blood pressure will be assessed using semiautomatic equipment, measuring systolic and diastolic pressures in millimeters of mercury (mmHg). Ambulatory Blood Pressure Monitoring (ABMP) will be employed at the beginning of the clinical trial. Lower readings indicate better blood pressure control, while higher readings suggest poorer control.
Increased Antihypertensive Medication Requirements in Patient Groups | From baseline (16th week) up to delivery
  The investigators will monitor both the inorganic nitrate group and the placebo group for any need to increase the dosage of antihypertensive medications, frequency or introduce a new agent.

SECONDARY OUTCOMES:
Doppler Analysis of Maternal and Fetal Vessel Behavior Across Pregnancy in Both Groups | From baseline (16th week) up to delivery
  Using Doppler velocimetry, the investigators will evaluate fetal vessels, focusing on the middle cerebral artery and umbilical artery. These tests will be conducted with mothers resting in left lateral decubitus during fetal rest periods, excluding respiratory movements. Key parameters, including the systole/diastole (A/B) ratios, resistance index, and pulsatility index, will be captured. Concurrently, maternal Doppler velocimetry of the uterine artery and pulse wave velocity will be measured to assess arterial stiffness.
Fetal Growth Assessment and Incidence of Fetal Growth Restriction in Both Groups | From baseline (16th week) up to delivery
  Fetal growth will be assessed using biometric measurements and evaluations like the fetal biophysical profile, placental maturity grade, and amniotic fluid evaluations. Key biometric parameters include biparietal diameter, cranial circumference, abdominal circumference, femur length, and estimated fetal weight (EFW). The "Hadlock" formula will help determine EFW, classifying the fetus as small for gestational age, average or large for gestational age. The biophysical profile will give insights into fetal movements and conditions over a 30-minute period. Placental maturity and amniotic fluid status will further provide context to the overall fetal health and growth.
Incidence of Preeclampsia Overlap and Adverse Maternal Outcomes in Each Group | At the time of delivery
  Clinical data will be collected to evaluate the presence of preeclampsia overlap and any associated adverse maternal outcomes. The collected data will include the gestational age at the time of delivery (in weeks + days), type of delivery (vaginal or cesarean), and specific clinical outcomes related to the mother's health
Incidence of Perinatal Outcomes | Immediately after delivery.
  Post childbirth, perinatal outcomes will be assessed by recording essential metrics of the newborn. The collected data will include the newborn's gender, weight (measured in grams), length (measured in cm), and the Apgar scores documented at both the first- and fifth minutes post-birth.
Vascular Reactivity of the Umbilical Artery In Vitro in Both Groups After Delivery | Approximately 15 to 30 minutes post-delivery, with some additional time for the in vitro evaluations.
  Umbilical cord fragments will b collected for evaluation. The fragments will be used to assess vascular tone changes in the umbilical artery using isometric force transducers. The viability and reactivity of the vessel rings will be determined using specific stimuli such as potassium chloride (KCl) and serotonin.
Evaluation of Complete Blood Count, Lipid and Glycemic Profiles, and Fasting Insulin Levels in Each Group | From baseline (16th week) up to delivery
  Participants' overall health will be evaluated through a series of blood tests, including complete blood count, glucose and insulin levels, creatinine, urea, liver enzymes, serum bilirubins and lipid profile.
Evaluation of Nitric Oxide Metabolite Concentrations in Plasma, Urine, and Saliva in Each Group | From baseline (16th week) up to delivery
  The concentrations of nitrate and nitrite, as key metabolites of nitric oxide, will be assessed in participants' plasma, urine, and saliva samples. The determination will be done using the Sievers Nitric Oxide Analyzer
Evaluation of Serum Markers for Preeclampsia in Each Group | From baseline (16th week) up to delivery
  The risk of developing preeclampsia will be assessed by calculating the soluble fms-like tyrosine kinase (sFLT-1) and placenta growth factor (PlGF) ratio using serum values of the angiogenic factors PlGF and sFLT-1. This ratio provides an indication of the likelihood of preeclampsia onset within specified time frames or the presence of placental insufficiency.
Evaluation of Inflammatory Markers in Each Group | From baseline (16th week) up to delivery
  Serum concentrations of various inflammatory markers, including adiponectin, intercellular adhesion molecule 1 (ICAM-1), interleukin-6 (IL6), interleukin-8 (IL8), interleukin-10 (IL10), leptin, resistin, tumor necrosis factor-alpha (TNFa), vascular cell adhesion molecule 1 (VCAM-1), vascular endothelial growth factor (VEGF), and visfatin, will be determined to evaluate inflammatory status in the participants.
Evaluation of Oxidative Stress Markers in Each Group | From baseline (16th week) up to delivery
  The extent of lipid peroxidation will be represented by plasma levels of malondialdehyde (MDA). Lower MDA levels suggest decreased oxidative damage. Simultaneously, the overall antioxidant activity in the plasma will be gauged through the ferric-reducing ability of plasma (FRAP). Elevated FRAP values indicate a heightened ability to resist oxidative stress.
Evaluation of Matrix Metalloproteinases and Inhibitors in Each Group | From baseline (16th week) up to delivery
  Serum concentrations of matrix metalloproteinases (MMPs) 2 and 9, as well as their inhibitors tissue inhibitor of metalloproteinases (TIMPs) 1 through 4, will be determined.
Evaluation of Diet Quality in Each Group Using the SISVAN Protocol | The SISVAN protocol will be employed at the enrollment.
  The quality of participants' diets will be assessed using a standardized SISVAN protocol. Concurrently, dietary recalls will be employed to provide a detailed account of participants' food consumption and nutritional patterns.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo C Cavalli, Dr, Principal Investigator — Medical School of Ribeirao Preto, USP
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto - USP, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No